CLINICAL TRIAL: NCT07102693
Title: Left Atrial Strain Assessment in Ischemic Stroke Patients: a Retrospective Case-control Study - the ASSISTANT Study
Brief Title: Left Atrial Strain Assessment in Ischemic Stroke Patients
Acronym: ASSISTANT
Status: Completed | Type: Observational
Sponsor: Connolly Hospital Blanchardstown (Other)
Responsible Party: Principal Investigator, Michael J Daly, MA MD PhD, Principal Investigator, Connolly Hospital Blanchardstown
Other Study IDs: CBH 024/23
Record Dates: First submitted 2025-07-30; First posted 2025-08-05 (Actual); Last update posted 2025-08-12 (Actual); Status verified 2025-08

CONDITIONS: Ischemic Stroke; Left Atrial Strain; Sinus Rhythm
Keywords: left atrial strain
MeSH Terms: conditions — Ischemic Stroke

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Retrospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- Patients with Acute Ischemic Stroke: Patients presenting to the emergency department with FAST positive symptoms who are proven to have acute ischaemic stroke on neuroimaging.
- Patients without Acute Ischaemic Stroke: Patients presenting to the emergency department with FAST positive symptoms who do not have evidence of acute ischaemic stroke on neuroimaging and an alternative cause of their FAST symptoms is found

SUMMARY:
This study is investigating a potential link between a novel measurement made on cardiac ultrasound and the risk of ischemic stroke in patients with a normal heart rhythm. The novel measurement is called left atrial strain. It uses speckle tracking echocardiography to measure the muscle function of the left atrium, one of the cardiac chambers. Investigators investigated whether patients with lower function of this chamber are at a higher risk of developing stroke from blood clots traveling to the brain. It is already known that patients with an irregular heart rhythm known as atrial fibrillation are at higher risk of these types of strokes. Investigators wanted to determine if there is a similar association in patients with normal heart rhythm but low left atrial strain.

ELIGIBILITY:
Inclusion Criteria:

* Emergency department presentation with FAST positive symptoms
* Neuroimaging performed as part of stroke workup
* Echocardiogram performed during index admission

Exclusion Criteria:

* Any history of atrial fibrillation prior or during admission
* Age below 18 years of age
* No echocardiogram or echocardiogram images not of sufficient quality to perform left atrial strain analysis
* At least moderate mitral regurgitation
* ASD or PFO

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients presenting to the emergency department with FAST positive symptoms suspicious for an acute stroke.
Sampling Method: Non-Probability Sample
Enrollment: 468 (Actual)
Dates: Start 2024-07-15 (Actual); Primary Completion 2025-06-01 (Actual); Study Completion 2025-06-01 (Actual)

PRIMARY OUTCOMES:
Correlation between left atrial strain and acute ischaemic stroke | 2 weeks
  This correlation will be adjusted for common stroke risk factors such as age, gender, hypertension, smoking, dyslipidaemia, and diabetes.

CONTACTS AND LOCATIONS:
Locations (1):
- Connolly Hospital Blanchardstown, Dublin, Co. Dublin, Ireland

IPD SHARING:
Plan to Share IPD: Yes
Echo measurements: Left atrial strain measurements, left ventricular ejection fraction, interventricular septal thickness, E/e' Demographics: Age, gender, hypertension status, smoking status, diabetes status, dyslipidaemia status,